CLINICAL TRIAL: NCT01060280
Title: The Effectiveness of the Physiotherapy Techniques Group GDS and Individual GDS for the Treatment of Nonspecific Low Back Pain in Primary Care. A Cluster, Randomized, Controlled Trial.
Brief Title: Effectiveness of Group GDS and Individual GDS for Treatment of Low Back Pain in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kovacs Foundation (Other)
Responsible Party: Principal Investigator, Francisco M. Kovacs, Director of Scientific Department, Kovacs Foundation, Kovacs Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FK-DO 30; FK-DO 10/020 (Other: Hospital Doce de Octubre, Madrid, Spain)
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Subacute Nonspecific Low Back Pain; Chronic Nonspecific Low Back Pain
Keywords: low back pain; physiotherapy; exercise; active management
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Education group (Active Comparator): Routine clinical practice (includes usual physiotherapy)plus education on active management.
  Interventions: Behavioral: Education on active management; Other: Group GDS physiotherapy; Other: Individual GDS physiotherapy
- Group GDS physiotherapy (Active Comparator): Routine clinical practice (except usual physiotherapy, which is substituted for Group GDS)plus education on active management.
  Interventions: Other: Group GDS physiotherapy; Other: Individual GDS physiotherapy
- Individual GDS physiotherapy (Active Comparator): Routine clinical practice (except for usual physiotherapy, which will be substituted by Group and Individual GDS) plus education on active management.
  Interventions: Other: Individual GDS physiotherapy

INTERVENTIONS:
Behavioral: Education on active management — Routine clinical practice plus education on active management.
  Arms: Education group
Other: Group GDS physiotherapy — Routine clinical practice (which will be substituted by Group GDS) plus education on active management.
  Arms: Education group; Group GDS physiotherapy
Other: Individual GDS physiotherapy — Routine clinical practice (except for usual physiotherapy, which is substituted by Group and Individual GDS) plus education on active management.

SUMMARY:
A cluster, randomized, controlled clinical trial, where the hypothesis is that Group GDS and Individual GDS are effective in the treatment of nonspecific low back pain. The clusters will be the participating physiotherapy departments in primary care who treat patients with low back pain. In each physiotherapy department there will be 3 groups: education group, Group GDS and Individual GDS. Patients will be followed for 12 months. Variables will be: demographic,intensity of pain, disability, quality of life, patient satisfaction, medication intake for current episode, non-pharmacologic treatment for current episode, co-morbidity, diagnostic tests, sick leave, and habitual physical activity. The questionnaires to be used are: Roland Morris Disability Questionnaire, PI-NRS, VAS, SF-12 and EQ-5d.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with nonspecific low back pain by the primary care physician
* more than or equal to 18 and less than or equal to 65 years of age

Exclusion Criteria:

* not signing the informed consent form
* pregnancy
* diagnosis of inflammatory rheumatologic disease, cancer, or fibromyalgia
* signs for suspicion of fibromyalgia
* having red flags for systemic disease
* presenting criteria for urgent referral to surgery
* presenting criteria for non-urgent referral to surgery
* inability to read, understand, or follow verbal orders (dementia,blindness, doesn´t know how to read)
* bedridden
* having received physiotherapy in last 12 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2010-05; Primary Completion 2011-10 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Low back pain, referred pain and disability | Baseline, 2, 6 and 12 months

SECONDARY OUTCOMES:
Self-reported health (PCS and MCS summaries of SF-12), and use of other pharmacologic and non-pharmacologic treatments | Baseline, 2, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Kovacs, MD, PhD, Study Director — Kovacs Foundation, Palma de Mallorca, Spain; Mario Gestoso, MD, Principal Investigator — Kovacs Foundation, Palma de Mallorca, Spain
Locations (1):
- Areas Nº 1 and 11. Primary Care. Spanish National Health Service in Madrid (SERMAS), Madrid, Madrid, Spain

REFERENCES:
- [Background] Frost H, Lamb SE, Doll HA, Carver PT, Stewart-Brown S. Randomised controlled trial of physiotherapy compared with advice for low back pain. BMJ. 2004 Sep 25;329(7468):708. doi: 10.1136/bmj.38216.868808.7C. Epub 2004 Sep 17. PMID 15377573
- [Background] Rivero-Arias O, Gray A, Frost H, Lamb SE, Stewart-Brown S. Cost-utility analysis of physiotherapy treatment compared with physiotherapy advice in low back pain. Spine (Phila Pa 1976). 2006 May 20;31(12):1381-7. doi: 10.1097/01.brs.0000218486.13659.d5. PMID 16721304
- [Background] Little P, Lewith G, Webley F, Evans M, Beattie A, Middleton K, Barnett J, Ballard K, Oxford F, Smith P, Yardley L, Hollinghurst S, Sharp D. Randomised controlled trial of Alexander technique lessons, exercise, and massage (ATEAM) for chronic and recurrent back pain. BMJ. 2008 Aug 19;337:a884. doi: 10.1136/bmj.a884. PMID 18713809
- [Derived] Diaz-Arribas MJ, Kovacs FM, Royuela A, Fernandez-Serrano M, Gutierrez-Fernandez L, San Martin-Pariente O, Abraira V, Ramos-Sanchez M, Llorca-Palomera R, Pardo-Hervas P, Gestoso M, Sanchez-Gil GC, Elena-Lucas MA, Paniagua-de-la-Calle R, Castellanos-Lopez I, Garcia-Heredia MA, Ceron-Sanz AM, Victoria-Gonzalez B, Monsalve-Martin C, Duque-Heras JM, Juanes-Hernandez MJ, Saura-Conti J, Soto-Saez JL, Roman-Moraleda C, Ruiz-Arias C, Martin-Mora B, Escolano-Garcia R, Cantero-Bengoechea JS, Garcia-Lopez E, Lopez-Pelegrin A, Padilla-Martin E, Martinez-Rodriguez M, Casillas-Martin J, Jerez-Vazquez J, Barrientos-Gomez L; Spanish Back Pain Research Network. Effectiveness of the Godelieve Denys-Struyf (GDS) method in people with low back pain: cluster randomized controlled trial. Phys Ther. 2015 Mar;95(3):319-36. doi: 10.2522/ptj.20140099. Epub 2014 Oct 30. PMID 25359444